CLINICAL TRIAL: NCT05479032
Title: Amantadine for Neuroenhancement in Acute Patients Study - A Prospective Pilot Proof of Concept Phase IIb Study in Intensive and Intermediate Care Unit Patients
Brief Title: Amantadine for Neuroenhancement in Acute Patients Study
Acronym: ANNES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-10
Record Dates: First submitted 2022-06-24; First posted 2022-07-28 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-02

CONDITIONS: Disorder of Consciousness
Keywords: Amantadine; Neuroenhancement
MeSH Terms: conditions — Consciousness Disorders | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Intensive care patients suffering from reduced consciousness not otherwise explained treated with Amantadine
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — 2x100 mg Amantadine for 3-5 days (dosage can be doubled in case of missing response to treatment after 48 hours)

SUMMARY:
Introduction: Many patients on intermediate care (IMC) and intensive care units (ICU) suffer from reduced consciousness. In this situation, a treatment attempt with Amantadine is often undertaken. While clinicians report good results with this approach, the treatment is off-label and the scientific evidence limited.

Study design: Monocenter, phase IIb, proof of concept, open-label pilot study. Methods: 50 intensive care patients with reduced consciousness not otherwise explained will be treated with Amantadine for 5 days. Vigilance is checked before, during and after treatment (on discharge and after 3 months) using electroencephalography (EEG) and established clinical tests, for instance Glasgow Coma Scale (GCS), Glasgow Outcome Scale - Extended (GOS-E), Coma Recovery Scale Revised (CRS-R) and others.

Results: The primary endpoint "improvement of the GCS scale from screening to day 5 of at least 3 points" is analysed according to the Simon design. The secondary endpoints (GCS continuous scale, modified Rankins Scale (mRS), National Institute of Health Stroke Scale (NIHSS), GOS-E, CRS-R and Montreal Cognitive Assessment (MoCA) after 90 days, Richmond Agitation-Sedation Scale (RASS) and Intensive Care Delirium Screening Checklist (ICDSC) will be analysed by mixed models with time (categorically coded) as only factor including all measurements up to 3 months follow up.

Discussion: The investigators aim to shed light on an established clinical practice without sufficient scientific evidence. The investigators are aware that the power of our study is limited by design (no control group, no blinding). However, if successful, this study may be the basis for a randomized controlled trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years at the time of signing the informed consent.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures or informed consent is signed
* As subject has per definition reduced consciousness and therefore is not in a position to provide written informed consent, inclusion of this patient is possible if the patient will give basic informed consent seven days after enrollment. Alternatively, the patient's relatives can give written informed consent.
* Able to adhere to the study visit schedule and other protocol requirements.
* Subject (male or female) is willing to use highly effective methods during treatment and for 4 days (male or female) after the end of treatment (adequate: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner1, sexual abstinence2).

  1. Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success
  2. In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
* All subjects must agree not to share medication.
* Reduced consciousness, defined as GCS <8, not otherwise explained
* Inconspicuous EEG and ECG

Exclusion Criteria:

* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials or observation period of competing trials.
* Age < 18 years
* Reduced consciousness, otherwise sufficiently explained
* Delirium (Intensive Care Delirium Screening Checklist (ICDSC) > 4 or >5 in aphasic patients)
* History of epileptic seizures or status epilepticus
* Pre-existing cardial conditions (e.g. heart failure (NYHA IV), cardiomyopathy, myocarditis, arrythmia (patients with a QTc time increase of >60ms or interval of >480ms have to be excluded from treatment), simultaneous treatment with other QT time elongating drugs, hypo-magnesaemia or -kalemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of vigilance measured by change in the Glasgow Coma Scale (GCS); a patient is defined as responder if his/her score increases by at least 3 points. | Assessment will take place before treatment (baseline value) and after 120 hours after treatment begin.
  The Glasgow Coma Scale (GCS) (Teasdale and Jennett, 1974) is a clinical scale used to measure a patient's level of consciousness. The GCS assesses patients based on their ability to perform limb and eye movements as well as to speak. These three categories represent the core elements of the scale: "eye", "verbal", and "motor". A person's GCS score can range from 3 (completely unresponsive) to 15 (completely responsive). This score is fast, easily and reliably to perform and can be used in emergency situations and also to monitor hospitalized patients.

SECONDARY OUTCOMES:
Change in vigilance reflected by change in the Richmond Agitation-Sedation Scale (RASS) | Assessment will take place before treatment (baseline value) and after 3 months.
  The Richmond Agitation Sedation Scale is a ten-step scale for assessment and quantification of sedation as well as agitation with the value '0' describing the physiological state, a value of '-5' deep sedation and '+4' severe agitation (Sessler et al., 2001).
Change of vigilance measured by the Full Outline of UnResponsive (FOUR) score | Assessment will take place before treatment (baseline value) and after 3 months.
  The FOUR Score is a clinical grading scale for the assessment of patients with an impaired level of consciousness. "FOUR" is an acronym for "Full Outline of UnResponsiveness". It is a 17-point scale with potential scores ranging from 0-16 (decreasing score associated with a worsening level of consciousness). The FOUR score overcomes some of the shortcomings of the GCS by assessing the four domains of neurological function: eye responses, motor responses, brainstem reflexes, and even breathing pattern (Wijdicks et al., 2005).
Appearance of delirium measured by change in the Intensive Care Delirium Screening Checklist (ICDSC) | Assessment will take place before treatment (baseline value) and after 3 months.
  The Intensive Care Delirium Screening Checklist can easily and quickly be applied by a clinician or a nurse in the critical care setting to screen all patients for a delirium (even when communication is compromised in case of aphasia). A value of 4 or more points corresponds with delirium. (Bergeron et al., 2001)
Change in symptoms measured by the National Institute of health Stroke Scale (NIHSS) | Assessment will take place before treatment (baseline value) and after 3 months.
  The National Institutes of Health Stroke Scale (NIHSS) is used to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability be-tween 0 and 4. For each item, a score of 0 indicates normal function, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (NIH, National Institute of Neurological Disorders and Stroke. https://www.ninds.nih.gov/sites/default/files/NIH_Stroke_Scale_Booklet.pdf).
Change in symptoms measured by the modified Rankin Scale (mRS) | Assessment will take place before treatment (baseline value) and after 3 months.
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It ranges from 0 (no symptoms) to 6 (death). (Wilson et al., 2002)
Change of vigilance measured by the Glasgow Outcome Scale - Extended (GOS-E) | Assessment will take place before treatment (baseline value) and after 3 months.
  The Glasgow Outcome Score (GOS) is a scale for patients with brain injuries, such as cerebral traumas or strokes that groups the victims by the objective degree of recovery (Jennett, 1975). Later, the same authors proposed to split the 3 better categories (severe disability to good recovery, i.e. 3 to 5) in lower and upper sub-categories, leading to the extended version of the scale (GOS-E) which includes 6 plus 2 (death and vegetative state), i.e. 8 categories in total (Jennett et al., 1981).
Change of vigilance measured by the Coma Recovery Scale revised (CRS-R) | Assessment will take place before treatment (baseline value) and after 3 months.
  The Coma Recovery Scale - Revised (CRS-R) is a standardized neurobehavioral assessment instrument for the usage in patients with disorders of consciousness. It is intended to establish diagnosis, monitor recovery, predict outcome as well as assess treatment effectiveness. A low score reflects reflexive activity, while a high score mirrors cognitively-mediated behaviors (Giacino et al., 2004)
Change of vigilance measured by the Montreal Cognitive Assessment (MoCA) | Assessment will take place before treatment (baseline value) and after 3 months.
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment (Nasreddine et al., 2005). It was validated in the setting of mild cognitive impairment, and has subsequently been adopted in numerous other clinical settings. A high score corresponds to high cognitive functioning.
Survival | Assessment will take place before treatment (baseline value) and after 3 months.
  Mortality
Change of vigilance measured by EEG (ratio of fast and slow oscillations) | Assessment will take place before treatment (baseline value) and after 3 months.
  A regular EEG will be recorded regularly as part of our routine clinical procedures in patients with reduced vigilance. Reduced vigilance is typically reflected by slow oscillations like delta or theta, thus vigilance will be measured by ratio between fast oscillations (alpha, beta) and slow oscillations (theta, delta).
Clinical change measured by the therapists' questionnaire | Assessment will take place before treatment (baseline value) and after 3 months.
  Therapists' questionnaire: This is a self-developed questionnaire for nursing staff as well as physiotherapists to even capture and assess the subtle clinical changes that might escape the standard scales within this heterogenous patient cohort. The seven items investigated mainly cover the patients' ability to - even at a very low level - interact with his/her environment and take part in e.g. physiotherapeutic procedures. Its total score ranges from 0 (best) to 21 (worst) points.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Feil, attending physician, Principal Investigator — University Hospital Tübingen, Deparment for Neurology and Stroke; Annerose Mengel, attending physician, Principal Investigator — University Hospital Tübingen, Deparment for Neurology and Stroke
Locations (1):
- Universitätsklinikum Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arciniegas DB, Frey KL, Anderson CA, Brousseau KM, Harris SN. Amantadine for neurobehavioural deficits following delayed post-hypoxic encephalopathy. Brain Inj. 2004 Dec;18(12):1309-18. doi: 10.1080/02699050410001720130. PMID 15666573
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Brioschi A, Gramigna S, Werth E, Staub F, Ruffieux C, Bassetti C, Schluep M, Annoni JM. Effect of modafinil on subjective fatigue in multiple sclerosis and stroke patients. Eur Neurol. 2009;62(4):243-9. doi: 10.1159/000232927. Epub 2009 Aug 7. PMID 19672078
- [Background] Clarencon F, Bardinet E, Martinerie J, Pelbarg V, Menjot de Champfleur N, Gupta R, Tollard E, Soto-Ares G, Ibarrola D, Schmitt E, Tourdias T, Degos V, Yelnik J, Dormont D, Puybasset L, Galanaud D; Neuro Imaging for Coma Emergence and Recovery (NICER) consortium. Lesions in deep gray nuclei after severe traumatic brain injury predict neurologic outcome. PLoS One. 2017 Nov 2;12(11):e0186641. doi: 10.1371/journal.pone.0186641. eCollection 2017. PMID 29095850
- [Background] DGN and AWMF (2016). S3-Leitlinie "Idiopathisches Parkinson-Syndrom". AWMF-Register-Nummer: 030-010. 2016.
- [Background] DGPPN, et al. (2016). S3-Leitlinie
- [Background] Gagnon DJ, Leclerc AM, Riker RR, Brown CS, May T, Nocella K, Cote J, Eldridge A, Seder DB. Amantadine and Modafinil as Neurostimulants During Post-stroke Care: A Systematic Review. Neurocrit Care. 2020 Aug;33(1):283-297. doi: 10.1007/s12028-020-00977-5. PMID 32394130
- [Background] Ghalaenovi H, Fattahi A, Koohpayehzadeh J, Khodadost M, Fatahi N, Taheri M, Azimi A, Rohani S, Rahatlou H. The effects of amantadine on traumatic brain injury outcome: a double-blind, randomized, controlled, clinical trial. Brain Inj. 2018;32(8):1050-1055. doi: 10.1080/02699052.2018.1476733. Epub 2018 May 23. PMID 29790790
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Gower A, Tiberi M. The Intersection of Central Dopamine System and Stroke: Potential Avenues Aiming at Enhancement of Motor Recovery. Front Synaptic Neurosci. 2018 Jul 6;10:18. doi: 10.3389/fnsyn.2018.00018. eCollection 2018. PMID 30034335
- [Background] Gualtieri T, Chandler M, Coons TB, Brown LT. Amantadine: a new clinical profile for traumatic brain injury. Clin Neuropharmacol. 1989 Aug;12(4):258-70. No abstract available. PMID 2680078
- [Background] Hubsher G, Haider M, Okun MS. Amantadine: the journey from fighting flu to treating Parkinson disease. Neurology. 2012 Apr 3;78(14):1096-9. doi: 10.1212/WNL.0b013e31824e8f0d. PMID 22474298
- [Background] Jang SH, Chang CH, Jung YJ, Kim JH, Kwon YH. Relationship Between Impaired Consciousness and Injury of Ascending Reticular Activating System in Patients With Intracerebral Hemorrhage. Stroke. 2019 Aug;50(8):2234-2237. doi: 10.1161/STROKEAHA.118.023710. Epub 2019 Jun 11. PMID 31181997
- [Background] Jang SH, Kim HS. Aneurysmal subarachnoid hemorrhage causes injury of the ascending reticular activating system: relation to consciousness. AJNR Am J Neuroradiol. 2015 Apr;36(4):667-71. doi: 10.3174/ajnr.A4203. Epub 2015 Jan 8. PMID 25572950
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Jennett B, Snoek J, Bond MR, Brooks N. Disability after severe head injury: observations on the use of the Glasgow Outcome Scale. J Neurol Neurosurg Psychiatry. 1981 Apr;44(4):285-93. doi: 10.1136/jnnp.44.4.285. PMID 6453957
- [Background] Jibiki, I., K. Morikawa, and N. Yamaguchi.
- [Background] Landucci E, Filippi L, Gerace E, Catarzi S, Guerrini R, Pellegrini-Giampietro DE. Neuroprotective effects of topiramate and memantine in combination with hypothermia in hypoxic-ischemic brain injury in vitro and in vivo. Neurosci Lett. 2018 Mar 6;668:103-107. doi: 10.1016/j.neulet.2018.01.023. Epub 2018 Jan 12. PMID 29339173
- [Background] Leclerc AM, Riker RR, Brown CS, May T, Nocella K, Cote J, Eldridge A, Seder DB, Gagnon DJ. Amantadine and Modafinil as Neurostimulants Following Acute Stroke: A Retrospective Study of Intensive Care Unit Patients. Neurocrit Care. 2021 Feb;34(1):102-111. doi: 10.1007/s12028-020-00986-4. PMID 32435964
- [Background] Li J, Zhang P, Wu S, Yuan R, Liu J, Tao W, Wang D, Liu M. Impaired consciousness at stroke onset in large hemisphere infarction: incidence, risk factors and outcome. Sci Rep. 2020 Aug 5;10(1):13170. doi: 10.1038/s41598-020-70172-1. PMID 32759986
- [Background] Lutkenhoff ES, Chiang J, Tshibanda L, Kamau E, Kirsch M, Pickard JD, Laureys S, Owen AM, Monti MM. Thalamic and extrathalamic mechanisms of consciousness after severe brain injury. Ann Neurol. 2015 Jul;78(1):68-76. doi: 10.1002/ana.24423. Epub 2015 May 4. PMID 25893530
- [Background] Meythaler JM, Brunner RC, Johnson A, Novack TA. Amantadine to improve neurorecovery in traumatic brain injury-associated diffuse axonal injury: a pilot double-blind randomized trial. J Head Trauma Rehabil. 2002 Aug;17(4):300-13. doi: 10.1097/00001199-200208000-00004. PMID 12105999
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] ratiopharm (2018). Fachinformation Amantadin-ratiopharm®200 mg Infusionslösung.
- [Background] Reznik ME, Yaghi S, Jayaraman MV, McTaggart RA, Hemendinger M, Mac Grory B, Burton TM, Cutting SM, Thompson BB, Wendell LC, Mahta A, Potter NS, Daiello LA, Kosar CM, Jones RN, Furie KL. Level of consciousness at discharge and associations with outcome after ischemic stroke. J Neurol Sci. 2018 Jul 15;390:102-107. doi: 10.1016/j.jns.2018.04.022. Epub 2018 Apr 14. PMID 29801867
- [Background] Rohaut B, Doyle KW, Reynolds AS, Igwe K, Couch C, Matory A, Rizvi B, Roh D, Velazquez A, Megjhani M, Park S, Agarwal S, Mauro CM, Li G, Eliseyev A, Perlbarg V, Connolly S, Brickman AM, Claassen J. Deep structural brain lesions associated with consciousness impairment early after hemorrhagic stroke. Sci Rep. 2019 Mar 12;9(1):4174. doi: 10.1038/s41598-019-41042-2. PMID 30862910
- [Background] Sessler CN, Grap MJ, Brophy GM. Multidisciplinary management of sedation and analgesia in critical care. Semin Respir Crit Care Med. 2001;22(2):211-26. doi: 10.1055/s-2001-13834. PMID 16088675
- [Background] Stinton C, McKeith I, Taylor JP, Lafortune L, Mioshi E, Mak E, Cambridge V, Mason J, Thomas A, O'Brien JT. Pharmacological Management of Lewy Body Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2015 Aug 1;172(8):731-42. doi: 10.1176/appi.ajp.2015.14121582. Epub 2015 Jun 18. PMID 26085043
- [Background] Suarez JI, Tarr RW, Selman WR. Aneurysmal subarachnoid hemorrhage. N Engl J Med. 2006 Jan 26;354(4):387-96. doi: 10.1056/NEJMra052732. No abstract available. PMID 16436770
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024
- [Background] Wilson JT, Hareendran A, Grant M, Baird T, Schulz UG, Muir KW, Bone I. Improving the assessment of outcomes in stroke: use of a structured interview to assign grades on the modified Rankin Scale. Stroke. 2002 Sep;33(9):2243-6. doi: 10.1161/01.str.0000027437.22450.bd. PMID 12215594
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Young GB. Coma. Ann N Y Acad Sci. 2009 Mar;1157:32-47. doi: 10.1111/j.1749-6632.2009.04471.x. PMID 19351354
- [Derived] Hofmann A, Blum C, Single C, Adeyemi K, Schwarz P, Siokas V, Rattay TW, Haberle HA, Riessen R, Brendel B, Haug I, Bosel R, Zago M, Martus P, Ziemann U, Mengel A, Feil K. Amantadine for NeuroenhaNcement in acutE patients Study - a protocol for a prospective pilot proof of concept phase IIb study in intensive and intermediate care unit patients (ANNES). BMC Neurol. 2023 Aug 22;23(1):308. doi: 10.1186/s12883-023-03345-w. PMID 37608315
- See also: Simon design calculator — http://linus.nci.nih.gov/cgi-bin/simonr/cgi_main